CLINICAL TRIAL: NCT00690456
Title: A Randomized, Double Blind, Placebo Controlled Study Evaluating the Glycemic Effect of Rimonabant Added to Metformin in Patients With Type 2 Diabetes Insufficiently Controlled With Metformin Monotherapy
Brief Title: Effect of Rimonabant and Metformin Combination on Glycemic Control in Patients With Type 2 Diabetes
Acronym: TOCCATA
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Company decision taken in light of demands by certain national health authorities
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EFC10518; 2007-004833-40 (EudraCT Number)
Record Dates: First submitted 2008-05-07; First posted 2008-06-04 (Estimated); Last update posted 2016-05-18 (Estimated); Status verified 2016-04

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Randomized Controlled Trial; Metformin
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Rimonabant; Metformin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Rimonabant (Experimental): Rimonabant 20 mg once daily on top of metformin
  Interventions: Drug: Rimonabant; Drug: Metformin
- Placebo (Placebo Comparator): Placebo (for Rimonabant) once daily on top of metformin
  Interventions: Drug: Placebo (for Rimonabant); Drug: Metformin

INTERVENTIONS:
Drug: Rimonabant — Tablet, oral administration
  Other Names: SR141716; Acomplia
  Arms: Rimonabant
Drug: Placebo (for Rimonabant) — Tablet, oral administration
  Arms: Placebo
Drug: Metformin — Metformin continued at stable dose as background therapy

SUMMARY:
The primary objective of the study is to determine the effect of rimonabant 20 mg daily when added to ongoing metformin therapy on glycemic control (HbA1c) over a 36 week period in patients with type 2 diabetes.

Secondary objectives include evaluation of other markers of glycemic control, lipid profile, body weight, and abdominal obesity. Also, the trial will study the safety of rimonabant when added to metformin over a period of 47 weeks.

DETAILED DESCRIPTION:
The total duration per patient will be approximately 49 weeks including a 36-week double-blind treatment period.

ELIGIBILITY:
Inclusion Criteria:

* History of type 2 diabetes
* HbA1c between 7% to 10% at screening visit
* Treatment with metformin only with a fixed and stable dose of 1500 mg/day or more for at least the past 3 months prior to screening visit

Exclusion Criteria:

* Within 3 months prior to screening visit: change in lipid modifying agent, administration of systemic corticosteroids for more than 10 days, use of any anti-obesity agent or drugs for weight loss
* Weight loss of more than 5 kg within 3 months prior to screening
* Administration of other investigational drugs within 30 days prior to screening visit
* Prior exposure to type 1 cannabinoid receptor (CB1) antagonists including rimonabant
* Presence or history of cancer within the past five years
* Pregnant or breast-feeding women
* Presence of any severe medical or psychological condition that, in the opinion of the investigator, would compromise the patient's safe participation including uncontrolled serious psychiatric illness such a major depression within the last 2 years, and history of other severe psychiatric disorders.

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 403 (Actual)
Dates: Start 2008-05; Primary Completion 2009-02 (Actual); Study Completion 2009-02 (Actual)

PRIMARY OUTCOMES:
Change from baseline in HbA1c | 36 weeks

SECONDARY OUTCOMES:
Change from baseline in fasting plasma glucose | 36 weeks
Change from baseline in body weight | 36 weeks
Percent change from baseline in HDL-C and Triglycerides | 36 weeks

CONTACTS AND LOCATIONS:
Overall Officials: ICD CSD, Study Director — Sanofi
Locations (13):
- Sanofi-Aventis Administrative Office, Bridgewater, New Jersey, United States
- Sanofi-Aventis Administrative Office, Jakarta, Indonesia
- Sanofi-Aventis Administrative Office, Vilnius, Lithuania
- Sanofi-Aventis Administrative Office, Kuala Lumpur, Malaysia
- Sanofi-Aventis Administrative Office, México, Mexico
- Sanofi-Aventis Administrative Office, Makati City, Philippines
- Sanofi-Aventis Administrative Office, Warsaw, Poland
- Sanofi-Aventis Administrative Office, Bucharest, Romania
- Sanofi-Aventis Administrative Office, Moscow, Russia
- Sanofi-Aventis Administrative Office, Brastislava, Slovakia
- Sanofi-Aventis Administrative Office, Taipei, Taiwan
- Sanofi-Aventis Administrative Office, Bangkok, Thailand
- Sanofi-Aventis Administrative Office, Kiev, Ukraine